CLINICAL TRIAL: NCT05882266
Title: The Role of Plant-Based Omega-3 Fatty Acids and Molecular Characterisation in Individuals with Cardiovascular(CVD) Risk At Beacon Hospital in Selangor
Brief Title: The Role of Plant-Based Omega-3 Fatty Acids and Molecular Characterisation in Individuals with Cardiovascular(CVD) Risk
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Collaborators: Beacon Hospital Sdn Bhd (Other)
Responsible Party: Principal Investigator, Gew Soon Peng, Principal Investigator, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RSCH ID-23-00839-PGP
Record Dates: First submitted 2023-04-24; First posted 2023-05-31 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Cardiovascular Risk
Keywords: cvd risk; cardiovascular risk; plant omega; plant based omega 3; omega 3

STUDY DESIGN:
Intervention Model Description: This is a non-weight loss interventional study. This study employed a single-blinded, randomised controlled, parallel design to compare the effect of plant-based omega-3 versus standard dietary therapy among individuals with CVD risk for 12 weeks. The randomisation will be done by an independent researcher. The intervention study had comprised two groups:
  * Treatment group: Receive standard dietary therapy and plant-based omega-3 supplemental beverage consumed once daily during breakfast.
  * Control group: Receive only standard dietary therapy
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The randomisation will be done by an independent researcher using block randomisation. No one except the independent researcher will know which group were assigned for each code. The file containing the info for each code will be kept by the independent researcher in Beacon Hospital.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): Receive standard dietary therapy and plant-based omega-3 supplemental beverage consumed once daily during breakfast.
  Interventions: Dietary Supplement: Plant Omega
- Control (Placebo Comparator): Receive only standard dietary therapy
  Interventions: Other: Dietary therapy only

INTERVENTIONS:
Dietary Supplement: Plant Omega — A commercial plant-based omega-3 beverage consumed once daily during breakfast
  Arms: Treatment
Other: Dietary therapy only — Standard dietary therapy
  Arms: Control

SUMMARY:
The goal of this clinical trial is to investigate the outcome of plant-based omega-3 intervention on lipid profile and blood pressure after 12 weeks and to study the molecular markers associated with the incidence of CVD risk. The main questions it aims to answer are:

* What is the role of plant-based omega-3 intervention on lipid profile and blood pressure of individuals with CVD risk after 12 weeks?
* What is the association between unique molecular markers and plant-based omega-3 intervention among individuals with CVD risk?

Participants will be subjected to two groups:

* Treatment group: Receive standard dietary therapy and plant-based omega-3 supplemental beverage consumed once daily during breakfast
* Control group: Receive only standard dietary therapy

Researcher will compare between treatment and control group to see the effect of plant based omega-3 on lipid profile and blood pressure after 12 weeks

DETAILED DESCRIPTION:
This study is a single-blinded, randomised controlled, parallel clinical trial with the aim to compare the effect of plant-based omega-3 versus standard dietary therapy among individuals with CVD risk for 12 weeks. The randomisation will be done by an independent researcher.

Following, the sample size for this study is 72 individuals with CVD risk, calculated based from two previous studies that investigated the effect of plant based omega 3 intake on cardiometabolic risk individuals and dairy beverages intake among type 2 diabetes mellitus patient.

Besides that, demographic information, medical history, medication history, social history, family history and nutritional information will be gathered using the Case Report Form (CRF) along with 3 days diet record and International Physical Activity Questionnaire (IPAQ) for physical activities assessment. Furthermore, anthropometric data, pain assessment, product sensory evaluation and compliance assessment will also be assessed using the same CRF form.

Correspondingly, 10-hour fasting blood sample (20ml) will be collected from a total of 72 subjects (treatment group, n=36 and control group, n= 36, respectively) for the blood test profiles and genotyping microarray analysis. Subjects need to avoid any alcohol intake, unusual amounts of physical activity and unusual amounts of food intake within 24-hour of blood taking. All the biochemical analyses will be done and entirely sponsored by Beacon Precision Diagnostics Sdn. Bhd. The study will be conducted in compliance with ethical principles outlined in the Declaration of Helsinki and Malaysian Good Clinical Practice Guideline.

Also, subjects shall be informed of the study during their usual clinic visits. They will be requested to contact investigators if they are interested. An appointment will be made where the subject information sheet will be provided and explained to them. If they are willing to participate, the consent forms will be signed and dated. If they need to, they are allowed to take the information sheet home to consult with their family members and another day for getting consent arranged. This study is an independent study, subjects can choose to withdraw at any time. Lastly, the investigators declare they have no conflict of interest.

ELIGIBILITY:
Inclusion Criteria:

* Malaysian aged 18 to 60 years
* BMI between 18.5 and 39.9 kg/m2
* Not on any weight loss therapy
* Is able to commit to 12 weeks of either intervention
* Presented signs of metabolic syndrome or moderate hypercholesterolemia

Exclusion Criteria:

* Those who are pregnant or lactating
* Had undergone bariatric surgery
* Who have acute illnesses such as flu
* Who has any diabetes-related chronic complications except hypertension and hyperlipidemia
* Having chronic diseases in particular cancer, liver, kidney, heart disease, stroke, or psychiatric illness
* Having eating disorder or hypothyroidism

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-12-20 (Estimated); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes in lipid profile after 12 weeks intervention of plant based omega 3 | Baseline and Week 12
  Changes in the lipid profile level of LDL, HDL, total cholesterol, triglyceride using standard metric (mmol/L)
Changes in the blood pressure after 12 weeks intervention of plant based omega 3 | Baseline and Week 12
  Changes in both systolic and diastolic blood pressure using the standard unit (mmHg)
Changes in microarray gene expression profile in blood from individual with CVD risk | Baseline and Week 12
  Changes in microarray gene expression profile in blood from individual with CVD risk, in response to the 12 weeks intake of plant based omega 3

SECONDARY OUTCOMES:
Changes in anti-inflammatory effect of plant-based omega-3 after 12 weeks | Baseline, Week 12
  Changes in high-sensitivity C-Reactive Protein (hs-CRP) using standard metric (mg/L)
Changes in fasting blood glucose after 12 weeks intervention of plant based omega-3 | Baseline, Week 12
  Changes in fasting blood glucose using standard metric (mmol/L)
Changes in glycated hemoglobin after 12 weeks intervention of plant based omega-3 | Baseline, Week 12
  Changes in glycated hemoglobin (hbA1c) using standard metric (%)
Changes in quality of life of individuals with CVD risk, before and after the consumption of plant-based omega 3 for 12 weeks | Baseline, Week 12
  Changes in pain score assess using the short 0-10 numeric pain scale. It is a validated self-reported instrument assessing average pain intensity over the past 24 hour period. Possible scores range from 0 (no pain) to 10 (worst possible pain).

CONTACTS AND LOCATIONS:
Overall Officials: Yoke Kqueen Cheah, Principal Investigator — Universiti Putra Malaysia
Locations (1):
- Beacon Hospital Sdn Bhd, Petaling Jaya, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schmidt KA, Cromer G, Burhans MS, Kuzma JN, Hagman DK, Fernando I, Murray M, Utzschneider KM, Holte S, Kraft J, Kratz M. The impact of diets rich in low-fat or full-fat dairy on glucose tolerance and its determinants: a randomized controlled trial. Am J Clin Nutr. 2021 Mar 11;113(3):534-547. doi: 10.1093/ajcn/nqaa301. PMID 33184632
- [Background] Tovar J, Nilsson A, Johansson M, Bjorck I. Combining functional features of whole-grain barley and legumes for dietary reduction of cardiometabolic risk: a randomised cross-over intervention in mature women. Br J Nutr. 2014 Feb;111(4):706-14. doi: 10.1017/S000711451300305X. Epub 2013 Sep 24. PMID 24063257